CLINICAL TRIAL: NCT05712642
Title: A Dosing Study of Two Different Doses (0.3125mg Versus 0.625mg) Intravitreal Bevacizumab for Type 1 ROP (Retinopathy of Prematurity)
Brief Title: A Dosing Study of Intravitreal Bevacizumab for Retinopathy of Prematurity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nooran Mohammed Abdelhameed Abdelkader, Assistant lecturer ophthalmology department Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-108-2019
Record Dates: First submitted 2023-01-17; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A recieved 0.3125mg intravitreal bevacizumab in both eyes (Experimental): 9 infants in group A with type 1 ROP , received 0.3125mg IVI of bevacizumab in both eyes, serum systemic levels of VEGF was measured at day 0 (before injection) , and 1 week and 4 weeks post injection .
  Interventions: Drug: Intravitreal Bevacizumab
- Group B received 0.625mg intravitreal bevacizumab in both eyes (Active Comparator): 10 infants in group B with type 1 ROP , received 0.625mg IVI of bevacizumab in both eyes, serum systemic levels of VEGF was measured at day 0 (before injection) , and 1 week and 4 weeks post injection .
  Interventions: Drug: Intravitreal Bevacizumab

INTERVENTIONS:
Drug: Intravitreal Bevacizumab — Serum systemic level of VEGF was measured before and after 1 week and 4 weeks of intravitreal injection of bevacizumab
  Other Names: Avastin

SUMMARY:
The aim of our study was to determine whether a low dose of 0.3125mg intravitreal bevacizumab is effective in treatment of type 1 ROP as the standard 0.625 mg dose., regarding :

Serum Systemic VEGF levels. Retinal Vascularization.

ELIGIBILITY:
Inclusion Criteria:

Infants with Type 1 ROP according to ETROP study which is defined as:

* Zone I ROP with plus disease
* Zone I, stage 3 ROP without plus disease
* Zone II, stage 2 or 3 ROP with plus disease

Exclusion Criteria:

* Eyes with previous intravitreal injection
* Eyes with previous laser therapy
* Eyes with any other intraocular pathology other than ROP (congenital cataract, congenital glaucoma, any retinal pathology other than ROP)

Ages: 28 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Change in the serum systemic VEGF pre- and post- intravitreal injection of bevacizumab in both groups. | at day 0 (baseline ) , 1 week and 4 weeks post-injection
  serum systemic VEGF measured using human VEGF ELISA kit
The number of infants without need for rescue therapy until 60 weeks of postmenstrual age after initial treatment. | "up to 60 weeks postmenstrual age"
  Rescue therapy is defined as the need of a second dose of 0.625 mg bevacizumab reinjection or laser at any time during follow up period.

SECONDARY OUTCOMES:
Occurrence of any adverse events from intravitreal-injection | Within 4 weeks from intravitreal injection
  endophthalmitis , retinal detachment , cataract , vitreous hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Nooran Abdelkader, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt